CLINICAL TRIAL: NCT04520971
Title: Closed-loop Insulin Delivery in Pregnant Women With Type 1 Diabetes: a Randomized Controlled Trial: the CRISTAL Study
Brief Title: Closed-loop Insulin Delivery in Pregnant Women With Type 1 Diabetes
Acronym: CRISTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Ghent (Other); Universitair Ziekenhuis Brussel (Other); University Hospital, Antwerp (Other); Imelda Hospital, Bonheiden (Other); AZ Sint-Jan AV (Other); AZ Delta (Other); Onze Lieve Vrouw Hospital (Other); General Hospital Groeninge (Other); AZ Nikolaas (Other); AZ Turnhout (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64308
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Type1 Diabetes
Keywords: closed-loop insulin delivery

STUDY DESIGN:
Intervention Model Description: 1/1 randomization to 780G or continue with standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 780G closed-loop (Experimental): 780 closed-loop insulin delivery system
  Interventions: Device: 780G
- standard of care (Active Comparator): standard of care treatment (continue with current treatment of insulin pump without closed-loop or multiple daily insulin injections).
  Interventions: Device: standard of care

INTERVENTIONS:
Device: 780G — 780G closed-loop insulin delivery system (Medtronic)
  Arms: 780G closed-loop
Device: standard of care — continue with standard of care treatment (pump without closed-loop or MDI)
  Arms: standard of care

SUMMARY:
Multi-centric open-label randomized controlled trial (RCT) with 11 Belgian centers and one Dutch center in pregnant women with type 1 diabetes to assess safety, efficacy, feasibility and cost-effectiveness of 780 MiniMed Medtronic hybrid closed-loop insulin system (intervention group) compared to standard of care therapy (control group).

DETAILED DESCRIPTION:
Women will be recruited with a singleton pregnancy up to 12 weeks gestation. Participants will be randomized 1/1 to 780 pump or standard of care (continue with current treatment of insulin pump without closed-loop or multiple daily insulin injections). Participants will be stratified according to study center, baseline Hba1c, and method of insulin delivery (pump or injections). Participants will be followed-up till delivery. To account for differences in the type of continuous glucose monitoring (CGM) used between the intervention group and the control group, the same CGM system as in the 780 insulin pump group (Guardian™ Sensor 3 and once available the Guardian 4 sensor) will be used in a blinded manner in the control group to collect CGM data during at least four different time points in pregnancy: at 14-17 weeks, 20-23 weeks, 26-29 weeks and 33-36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with type 1 diabetes (T1DM), diagnosed with T1DM at least 1 year before pregnancy
* Age 18-45 years
* A singleton pregnancy confirmed by b-HCG in blood and/or ultrasound-confirmed gestational age up to 11 weeks and 6 days.
* Treated with intensive insulin treatment (either MDI or insulin pump). A closed-loop system can only be used in manual mode.
* Have a booking HbA1c (measurement taken at the first antenatal clinic visit after confirmed pregnancy) level ≤10%.
* Participants need to speak and understand Flemish, French or English and have e-mail access.

Exclusion Criteria:

* The use of a closed-loop insulin delivery system in auto mode.
* A twin (multiple) pregnancy
* A physical or psychological disease likely to interfere with the conduct of the study (based on the evaluation by the treating physician)
* Medications known to interfere with glucose metabolism
* An insulin dose of ≥1.5 units/kg
* Known allergy to adhesives due to infusion set and/or CGM

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
time in range | from 14 weeks to 36 weeks
  time between 63-140mg/dl (pregnancy glycemic target range)

SECONDARY OUTCOMES:
time in range during the night | from 14 weeks to 36 weeks
  time in range (63-140mg/dl) from midnight till 6am
time below low day and night | from 14 weeks to 36 weeks
  time <63mg/dl day and night
overnight time low | from 14 weeks to 36 weeks
  time <63mg/dl from midnight till 6am
time in range during the day | from 14 weeks to 36 weeks
  time in range (63-140mg/dl) during the day
time in range early pregnancy | from 9 weeks to 12 weeks
  time in range (63-140mg/dl) 9-12 weeks
time in range during each trimester | from 9 weeks to 36 weeks
  time in range (63-140mg/dl) during each trimester
HbA1c during each trimester | from 9 weeks to 36 weeks
  HbA1c (% and mmol/mol) during each trimester
mean glucose | from 14 weeks to 36 weeks
  mean glucose based on CGM
time above target (140mg/dl) | from 14 weeks to 36 weeks
  time >140mg/dl
time above target (180mg/dl) | from 14 weeks to 36 weeks
  time >180mg/dl
time below target (50mg/dl) | from 14 weeks to 36 weeks
  time <50mg/dl
time below target (54mg/dl) | from 14 weeks to 36 weeks
  time <54mg/dl
duration of hypoglycemia | from 14 weeks to 36 weeks
  low blood glucose index
time in nonpregnant target range | from 14 weeks to 36 weeks
  time 70-180mg/dl
CGM compliance | from 14 weeks to 36 weeks
  % of time use of CGM
insulin dose | from 14 weeks to 36 weeks
  total insulin dose
glycemic variability | from 14 weeks to 36 weeks
  standard deviation glucose values based on CGM
variation glucose values | from 14 weeks to 36 weeks
  coefficient of variation based on CGM
MAGE (mean amplitude of glycemic excursions) | from 14 weeks to 36 weeks
  mean amplitude of glucose variations based on CGM
nocturnal hypoglycemia | from 9 weeks to 36 weeks
  glucose <50mg/dl from 23-07hour
severe hypoglycemia | from 9 weeks to 36 weeks
  hypoglycemia requiring third-part assistance
rate of diabetic keto-acidosis | from 9 weeks to 36 weeks
  metabolic keto-acidosis with decreased ph and/or decreased bicarbonate in blood
gestational duration | delivery
  duration of pregnancy (weeks)
duration hospitalization delivery | delivery
  length of hospital stay (days)
type of labor | delivery
  spontaneous, induced or cesarean section before labor
type of delivery | delivery
  vaginal, forceps or vacuum, cesarean section during labor or planned cesarean section
rate of preterm delivery | delivery
  delivery <37 weeks
rate of gestational hypertension | from 20 weeks to delivery
  blood pressure of 140/90 mmHg or higher starting after 20 weeks of gestation
rate of worsening of chronic hypertension | from 9 weeks to delivery
  blood pressure of 140/90 mmHg or higher start is present before 20 weeks of gestation
rate of preeclampsia | from 20 weeks to delivery
  onset of new hypertension and proteinuria and/or end-organ dysfunction after 20 weeks of gestation
rate of eclampsia | from 20 weeks to delivery
  generalized convulsions and/or coma
rate of HELLP syndrome | from 20 weeks to delivery
  hemolysis, elevated liver enzymes and a low platelet count
rate of IUGR (intra-uterine growth restriction) | from 20 weeks to delivery
  intra-uterine growth restriction
rate of fetal malformation | up to 24 weeks
  congenital malformation
rate of miscarriage | <20 weeks
  fetal loss <20 weeks gestations
rate of termination of pregnancy | up to 24 weeks
  induced abortion
rate of stillbirth | >20 weeks
  mors in utero >20 weeks
rate of neonatal death | 1 month after delivery
  death <1 months after delivery
sex of infant | delivery
  boy or girl
birth weight | delivery
  birth weight (Kg and g)
rate of shoulder dystocia | delivery
  one or both of a baby's shoulders get stuck inside the mother's pelvis during labor.
rate of birth trauma | delivery
  fracture, damage to nerves...
rate of respiratory distress | delivery
  respiratory failure or distress
rate of hyperbilirubinaemia | delivery
  hyperbilirubinaemia with need of treatment with phototherapy
rate of macrosomia | delivery
  birth weight >4 Kg
rate with high birth weight | delivery
  birth weight >4.5 Kg
rate of LGA infant (large for gestational age) | delivery
  gestational age adjusted birth weight >90th percentile according to the standardized Flemish birth charts adjusted for parity and sex
rate of SGA infant (small for gestational age) | delivery
  gestational age adjusted birth weight <10th percentile according to the standardized Flemish birth charts adjusted for parity and sex
number with very large gestational age infants | delivery
  gestational age adjusted birth weight >97th percentile according to the standardized Flemish birth charts adjusted for parity and sex
cord blood ph | delivery
  cord blood gas ph
rate of neonatal hypoglycemia | up to 5 days after delivery
  neonatal hypoglycemia requiring intravenous dextrose
rate of NICU admission | up to 30 days after delivery
  Neonatal intensive care unit (NICU) admission defined as requiring a duration of at least 24 h
duration NICU admission | up to 30 days after delivery
  duration of NICU admission (days or weeks)
rate of fetal hyperinsulinemia | delivery
  cord blood c-peptide
skinfolds newborn | up to 3 days after delivery
  sum of skinfolds (triceps, scapula and flank)
neonatal fat mass | up to 3 days after delivery
  fat mass calculated by the formula of Catalano et al.
number with composite neonatal outcome | delivery
  pregnancy loss (miscarriage, still birth or neonatal death), LGA (large for gestational age), respiratory distress syndrome, birth trauma, shoulder dystocia, neonatal hypoglycemia and NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Benhalima, MD PhD, Principal Investigator — UZ Leuven
Locations (12):
- Belgium (11):
  - OLV Aalst-Asse, Aalst, Oost-Vlaanderen
  - Imelda Bonheiden, Bonheiden
  - AZ St Jan Brugge, Bruges
  - UZ Brussel, Brussels
  - UCLouvain, Brussels
  - UZ Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - UZ Leuven, Leuven
  - AZ Roeselare, Roeselare
  - AZ Nikolaas, Sint-Niklaas
  - AZ Turnhout, Turnhout
- Amsterdam UMC, Amsterdam, Netherlands

REFERENCES:
- [Background] Beunen K, Van Wilder N, Ballaux D, Vanhaverbeke G, Taes Y, Aers XP, Nobels F, Marlier J, Lee D, Cuypers J, Preumont V, Siegelaar SE, Painter RC, Laenen A, Gillard P, Mathieu C, Benhalima K. Closed-loop insulin delivery in pregnant women with type 1 diabetes (CRISTAL): a multicentre randomized controlled trial - study protocol. BMC Pregnancy Childbirth. 2023 Mar 16;23(1):180. doi: 10.1186/s12884-023-05481-0. PMID 36927458
- [Result] Benhalima K, Beunen K, Van Wilder N, Ballaux D, Vanhaverbeke G, Taes Y, Aers XP, Nobels F, Marlier J, Lee D, Cuypers J, Preumont V, Siegelaar SE, Painter RC, Laenen A, Gillard P, Mathieu C. Comparing advanced hybrid closed loop therapy and standard insulin therapy in pregnant women with type 1 diabetes (CRISTAL): a parallel-group, open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2024 Jun;12(6):390-403. doi: 10.1016/S2213-8587(24)00089-5. Epub 2024 Apr 30. PMID 38697182